CLINICAL TRIAL: NCT03589690
Title: Assessment of the Effect of Alpha Lipoic Acid Supplementation on Inflammatory Factors, Insulin Resistance, Glycemic Control and Anthropometric Indices in Patients With Metabolic Syndrome
Brief Title: Alpha Lipoic Acid Supplementation and Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. B.Abbasi (Other)
Responsible Party: Sponsor-Investigator, Dr. B.Abbasi, Clinical Professor, Science & Research Islamic Azad University Branch Khozestan
Organization: Science & Research Islamic Azad University Branch Khozestan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.IAU.SRB.REC.1396.82
Record Dates: First submitted 2018-02-27; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Thioctic Acid; Inflammation; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Insulin Resistance | interventions — Thioctic Acid

STUDY DESIGN:
Intervention Model Description: In this study, samples will be randomly divided into two groups receiving the supplement or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be conducted as a parallel randomized double-blind clinical trial. patient will randomly be divided into two groups, each will receive supplement or placebo for 12 weeks .Before the study, containers will be coded as A and B by a person other than the study researchers according the concealment rules .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha Lipoic acid (Experimental): Alpha lipoic acid capsules (600 mg/day)
  Interventions: Dietary Supplement: Alpha lipoic acid
- Placebo (Placebo Comparator): Starch-filled capsules (600 mg/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha lipoic acid — 22 Patients will consume 600 mg Alpha lipoic acid for 12 weeks .
  Other Names: Thioctic acid , ALA (Alpha lipoic acid)
  Arms: Alpha Lipoic acid
Dietary Supplement: Placebo — Participants will be supplemented with 600 mg/day placebo (Starch).
  Arms: Placebo

SUMMARY:
Metabolic syndrome is a collection of metabolic disorders. Abdominal obesity, dyslipidemia, reduced levels of high-density lipoprotein cholesterol, increased levels of serum triglyceride, insulin resistance are among the risk factors for metabolic syndrome and it has a global prevalence of 10 - 50 %.

Alpha-lipoic acid or thioctic acid is an antioxidant that may have effects on inflammatory pathways, glucose control indicators, blood pressure, lipid profiles, body weight, fat mass, and food intake regulation.

This study will be conducted as a parallel randomized double-blind clinical trial. In this study, 44 patients will be enrolled from endocrine and metabolism center of Shariati Hospital where their metabolic syndrome was diagnosed by an endocrinologist. At the beginning of the study written a self -administration will be taken from all patients.

In this study, patient will be randomly divided into two groups, each will be received supplement or placebo for 12 weeks. 22 of patients will be consume 600 mg Alpha lipoic acid for 12 weeks and 22 of patients will be consume 600 mg placebo (starch-filled) capsules daily. Both supplementation and placebo are provided from "Sepehr Drug and Treatment" company. Before the study, containers will be coded as A and B by a person other than the study researchers according to concealment rules. Physical activity information will be collected using short-IPAQ (International Physical Activity Questionnaire) and demographic information through a general information questionnaire. In order to evaluate dietary intake of patients in terms of energy(kcal/(day), carbohydrate(gr/day), protein(gr/day), fat intake(gr/day), SFA (Saturated fatty acids) (gr/day), MUFA (Monounsaturated fatty acids) (gr/day), PUFA (Polyunsaturated fatty acids)(gr/day), Vitamin E(mg/day), Vitamin C(mg/day), Beta-carotene(mg/day) and Sodium intake (mg/day), 24-hr recalls will be completed by interviewing the patient for 3 days (two normal days and a weekend day). Weight will be measured with the minimum dress and without shoes by using a digital balance scale of 100 grams and height will be measured without shoes by meters mounted to the wall with an accuracy of 0.1 centimeters. Then the body mass index will be calculated by dividing the weight (kg) by the square of the height (m), waist circumference will be measured in the narrowest area between the lowest lumbar spine and the iliac bone (cm), systolic and diastolic blood pressure will be measured after 15 minutes of rest, twice using the mercuric barometric measure and the mean will be reported as individual blood pressure. The blood sample will be taken after 12 hours of overnight fasting in two groups for measuring fasting blood glucose(mg/dL), lipid profile(mg/dL), glycosylated hemoglobin(percentage), serum insulin concentration (uIU/ml) ,TAC (Total antioxidant capacity) (umol/L), CRP (C-reactive protein) (ng/ml) and TNF-a (Tumor necrosis factor-a ) (pg/ml)and will be used the HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) formula to determine insulin resistance. All these steps will be completed at the start and end of the study. At the end of the study, counting the remaining capsules, the patient's compliance rate will be evaluated, and patients who have not consumed less than 90% of their capsules will be excluded from the analysis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel clinical trial of lipoic acid for inflammatory factors, insulin resistance, glycemic control and anthropometric indices in patients with metabolic syndrome. patients are randomly shared into two groups and received 600 mg supplemental and placebo for 12 weeks, Then the body mass index, waist circumference, systolic and diastolic blood pressure, FBS (fasting blood sugar), lipid profile ,HbA1C, serum insulin concentration, TAC, CRP and TNF-a , Insulin resistance are measured ;All these steps will be done at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. having 3 criteria or more of the Metabolic Syndrome criteria presented in NCEP:ATP III (National Cholesterol Education Panel : Adult Treatment Panel III)
2. Adults(18-60 y)
3. PO (not fasting) and oral feeding ability
4. full person's willingness to cooperate in the project
5. Lack of digestive problems
6. Not pregnancy and Lactation
7. No history of myocardial infarction and brain stroke in the past year
8. Diabetes controlled
9. Lack of any Cardiovascular disease

Exclusion Criteria

1. Pregnancy
2. Cardiovascular and brain stroke
3. Diagnosis of uncontrolled diabetes during research
4. Have any need for medication that may interfere in the study process
5. Unwillingness to continue the cooperation of each research unit
6. Death of each research unit
7. Consume less than %90 of the number of supplement and placebo to be eaten
8. Involvement in other clinical trial in last three months
9. Menopause

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-07-25 (Estimated); Primary Completion 2019-04-25 (Estimated); Study Completion 2019-07-25 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of CRP | Baseline and 12 weeks after
  Serum C-reactive protein (ng/ml)

SECONDARY OUTCOMES:
Change from baseline of Tnf-a | Baseline and 12 weeks after
  Serum tumor necrosis factor-a (pg/ml)
Change from baseline of FBS | Baseline and 12 weeks after
  Fasting blood glucose concentration (mg/dl)
Change from baseline of Triglyceride | Baseline and 12 weeks after
  Serum TG (triacylglycerol) concentration (mg/dl)
Change from baseline of total cholesterol | Baseline and 12 weeks after
  Serum TC (total cholesterol) concentration (mg/dl)
Change from baseline of LDL-Cholesterol | Baseline and 12 weeks after
  Serum LDL concentration (mg/dl)

IPD SHARING:
Plan to Share IPD: No